CLINICAL TRIAL: NCT01121328
Title: Autologous Umbilical Cord Blood Transfusion for Preterm and Low Birth Weight Neonates: A Pilot Feasibility Study
Brief Title: Autologous Umbilical Cord Blood Transfusion for Preterm Neonates
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No recruitment
Sponsor: Sahar M.A. Hassanein, MD (Other)
Responsible Party: Sponsor-Investigator, Sahar M.A. Hassanein, MD, Professor of Pediatrics, Children's Hospital, Faculty of Medicine, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB#1
Record Dates: First submitted 2010-05-03; First posted 2010-05-12 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Prematurity; Respiratory Distress Syndrome; Anemia of Prematurity; Intraventricular Hemorrhage
Keywords: Preterm neonates.; Autologous cord blood transfusion.
MeSH Terms: conditions — Premature Birth; Respiratory Distress Syndrome; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Autologous cord blood transfusion (Experimental): Collected cord blood at birth will be transfused for the preterm neonate
  Interventions: Biological: Autologous cord blood transfusion for preterm neonates; Biological: Autologous cord blood transfusion

INTERVENTIONS:
Biological: Autologous cord blood transfusion for preterm neonates — Cord blood collection after delivery of the baby. Preservation of blood in blood bank. Transfusion of blood within the first 14 postnatal days to maintain Hb level above 10gm%.
  Other Names: Transfusion blood bag collection.
Biological: Autologous cord blood transfusion — After delivery of the baby and before placental delivery in vaginal delivery. After delivery of the baby the placental will be taken out in cesarean section. sterilization of the umbilical cord will be done. Puncture of the umbilical cord vein with the needle of blood transfusion bag will be done.
  Blood will be kept in the blood bank. Blood grouping, haematocrit and CBC will be done for the cord blood.Maternal sample will be analysed simultaneously.
  Mononuclear layer will be separated within 6 hours and transfused to the preterm neonate immediately.
  RBCs will be separated and kept till need (Hb less than 10 gm%).
  Other Names: Cord blood transfusion for preterm neonates

SUMMARY:
This is a pilot study to test feasibility of collection, preparation and infusion of a baby's own (autologous) umbilical cord blood in the first 14 days after birth if the baby is born premature <35 weeks of gestation.

DETAILED DESCRIPTION:
In Egypt, 12-15.8% of live neonates are low birth weight and it is estimated that about one third of such infants are preterm [1] (UNICEF, 2001). In a study that Campbell et al. (2004) conducted in Egypt, the neonatal mortality rate was estimated to be 25 per 1000 live births. prematurity was considered the main cause of neonatal deaths (39%), followed by asphyxia (18%), infection (7%), especially in the late neonatal period, and congenital malformations (6%). A substantial proportion (29%) could not be classified [2]. In developing countries, prematurity was the main cause of early neonatal deaths (62%)[3] Autologous cord blood transfusion will be safe, and cheap. The preterm neonates need transfusion of whole blood or any of its components at a time during NICU admission.

ELIGIBILITY:
Inclusion Criteria:

* Preterm neonates less than 34 weeks of gestation.
* Low birth weight less than 1500 grams

Exclusion Criteria:

* Congenital malformations.
* Suspected inborn error of metabolism.
* Suspected inherited neurologic disease.

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2011-07; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Duration of mechanical ventilation | 30 days
  -No need for mechanical ventilation.

SECONDARY OUTCOMES:
Survival | 18 months
  * Survival until 12 months of age.
  * Improved physical growth and weight gain.
  * Neurodevelopmental outcome at 6, 12 and 18 months of age.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Sahar MA Hassanein, MD, Principal Investigator — Children's Hospital, Faculty of Medicine, Ain Shams University
Locations (1):
- Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt